CLINICAL TRIAL: NCT01855828
Title: Single Arm, Neoadjuvant, Phase II Trial of Pertuzumab and Trastuzumab Administered Concomitantly With Weekly Paclitaxel and FEC for Clinical Stage I-II HER2-Positive Breast Cancer
Brief Title: Phase 2 Trial of Pertuzumab and Trastuzumab With Weekly Paclitaxel and Chemotherapy for HER2 Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1305012136
Record Dates: First submitted 2013-05-13; First posted 2013-05-17 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Her2-Positive Breast Cancer
MeSH Terms: interventions — pertuzumab; Trastuzumab; Paclitaxel; Fluorouracil; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemo plus Pertuzumab,Trastuzumab (Experimental): During weeks 1-12, patients will receive pertuzumab, trastuzumab, and paclitaxel at the same time; during weeks 13-24 patients will receive pertuzumab and trastuzumab at the same time with 5-fluorouracil, epirubicin, and cyclophosphamide (FEC).
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab; Drug: Paclitaxel; Drug: 5-fluorouracil; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pertuzumab — First dose is 840mg, maintenance dose is 420mg. Pertuzumab will be administered once every 3 weeks for 24 weeks (8 doses total)
  Other Names: Perjeta
Drug: Trastuzumab — For weeks 1-12, first dose is 4 mg/kg, maintenance dose is 2 mg/kg administered every week (12 doses total).
  For weeks 13-24, dose is 6mg/kg administered every 3 weeks (4 doses total).
  Other Names: Herceptin
Drug: Paclitaxel — Administered at 80mg/m2 every week from week 1 to 12 (12 doses total).
  Other Names: Taxol
Drug: 5-fluorouracil — Administered at 500 mg/m2 for every 3 weeks during weeks 13-24 (4 doses total).
  Other Names: 5-FU
Drug: Epirubicin — Administered at 75mg/m2 every 3 weeks during weeks 13-24 (4 doses total).
  Other Names: Ellence
Drug: Cyclophosphamide — Administered at 500mg/m2 for every 3 weeks during weeks 13-24 (4 doses total).
  Other Names: Cytoxan

SUMMARY:
The main goal of this clinical trial is to test if adding pertuzumab (Perjeta), improves the anticancer activity of the combination chemotherapy regimen of trastuzumab (Herceptin) concomitant with paclitaxel, 5-fluorouracil, epirubicin, and cyclophosphamide (T-FEC). The study will also test the safety of this therapy.

DETAILED DESCRIPTION:
Subjects will receive 6 months of T-FEC chemotherapy concomitant with trastuzumab and pertuzumab before surgery. Subsequently, subjects will undergo surgery to remove any cancer from the breast and axillary lymph nodes that may have survived the chemotherapy. It is expected that the majority of women will have no viable cancer left in the breast or lymph nodes by the time all chemotherapy is completed.

ELIGIBILITY:
Inclusion Criteria:

- Patients with histologically confirmed stage I-III, HER2-positive invasive breast cancer for which adjuvant/neoadjuvant chemotherapy is indicated based on physician judgment following NCCN practice guidelines.

HER2 overexpression or amplification will be based on local test results and is defined as either:

(i) IHC staining of 3+ (uniform, intense membrane staining) in greater than or equal to 10% of invasive tumor cells or, (ii) Fluorescent in situ hybridization (FISH) result of more than six HER2 gene copies per nucleus or, (iii) FISH ratio (HER2 gene signals to chromosome 17 signals) of greater than or equal to 2.0.

* Patients with synchronous bilateral breast cancers are eligible if at least one of the tumors is HER2-positive.
* Left Ventricular Ejection Fraction (LVEF) greater or equal to 50% at baseline as determined by either ECHO or MUGA, or within the institution's normal limits.
* Women of childbearing potential must have a negative pregnancy test (serum or urine beta HCG) prior to initiation of chemotherapy. Both female and male breast cancer patients who are sexually active have to agree to practice contraception while participating in the trial and for 3 month after completion of therapy.
* Adequate bone marrow function as indicated by the following:
* ANC greater than or equal to 1500/uL
* Platelets greater than or equal to 100,000/uL
* Hemoglobin greater than or equal to 10 g/dL
* Adequate renal function, as indicated by creatinine less than or equal to 1.5 times upper limit of normal (ULN)
* Adequate liver function, as indicated by bilirubin less than or equal to 1.5 X ULN and AST or ALT less than or equal to 2x ULN.
* Signed informed consent.

Exclusion Criteria:

Patients will be excluded from the study based on any of the following criteria:

* Patients who underwent partial excisional biopsy, lumpectomy, segmental mastectomy, modified radical mastectomy or sentinel node biopsy and, therefore cannot be assessed for pathologic response accurately.
* Patients who are high risk for developing the following anthracycline, paclitaxel, trastuzumab or pertuzumab related toxicities including:

History of congestive heart failure, myocardial infarction or cardiomyopathy, uncontrolled hypertension despite adequate medications Pre-existing peripheral neuropathy > grade 3 Prior anthracycline therapy Known hypersensitivity to any of the study medications Patients older than age 65 due to increased risk of cardiotoxicity

* Active infection requiring systemic antibiotic therapy.
* Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Pusztai, MD, Principal Investigator — Yale University
Locations (1):
- Yale University Smilow Cancer Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemo Plus Pertuzumab,Trastuzumab: During weeks 1-12, patients will receive pertuzumab, trastuzumab, and paclitaxel at the same time; during weeks 13-24 patients will receive pertuzumab and trastuzumab at the same time with 5-fluorouracil, epirubicin, and cyclophosphamide (FEC).
  Pertuzumab: First dose is 840mg, maintenance dose is 420mg. Pertuzumab will be administered once every 3 weeks for 24 weeks (8 doses total)
  Trastuzumab: For weeks 1-12, first dose is 4 mg/kg, maintenance dose is 2 mg/kg administered every week (12 doses total).
  For weeks 13-24, dose is 6mg/kg administered every 3 weeks (4 doses total).
  Paclitaxel: Administered at 80mg/m2 every week from week 1 to 12 (12 doses total).
  5-fluorouracil: Administered at 500 mg/m2 for every 3 weeks during weeks 13-24 (4 doses total).
  Epirubicin: Administered at 75mg/m2 every 3 weeks during weeks 13-24 (4 doses total).
  Cyclophosphamide: Administered at 500mg/m2 for every 3 weeks during weeks 13-24 (4 doses total).
Period: Overall Study
Arm/Group | Chemo Plus Pertuzumab,Trastuzumab
Started | 50
Completed | 48
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chemo Plus Pertuzumab,Trastuzumab
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 51 [24 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 36
  Race/Ethnicity: African American | 4
  Race/Ethnicity: Asian | 2
  Race/Ethnicity: Hispanic | 6
  Race/Ethnicity: Unknown | 2
Region of Enrollment [Number; unit: participants]
  United States | 50
Hormone receptor status [Count of Participants; unit: Participants] — Receptor status retrieved from the subjects diagnostic pathology report.
  Participants
    Estrogen Receptor + / Progesterone Receptor + | 20
    Estrogen Receptor + / Progesterone Receptor - | 4
    Estrogen Receptor - / Progesterone Receptor - | 26
HER2 status [Count of Participants; unit: Participants] — Fluorescence in situ hybridization (FISH) and Immunohistochemistry (IHC) are tests used to detect breast cancer genetically. A positive FISH test and ICH status of 3+ are markers of HER2 status. These data were retrieved from the subjects' diagnostic pathology report and demonstrate the manner in which these patients were diagnosed.
  Participants
    Fluorescence in situ hybridization (FISH) positive | 27
    Immunohistochemistry (IHC) 3+ | 23
Clinical Tumor Status [Count of Participants; unit: Participants] — Baseline clinical staging
  Participants
    T1: Tumor is 2 cm or smaller | 18
    T2: Tumor is larger than 2 cm, but no larger than | 25
    T3: Tumor is larger than 5 cm | 5
    T4: Tumor is any size, but has spread | 2
Type of surgery [Count of Participants; unit: Participants] — The type of surgery describes the manner in which the patients' breast cancer was addressed surgically.
  Participants
    Mastectomy | 35
    Breast conserving surgery | 13
    No surgery (dropped out of study) | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With a Pathologic Complete Response Rate
Description: To estimate the pathologic complete response rate (pCR) when pertuzumab is added to weekly trastuzumab/paclitaxel followed by trastuzumab/5-fluorouracil, epirubicin and cyclophosphamide neoadjuvant chemotherapy in HER2-positive breast cancer. This study will assess pCR rates separately in ER+ and ER- cancers. Pathologic complete response is defined as no evidence of viable invasive tumor cells at the primary tumor site and axillary lymph nodes in the surgical specimen. Residual Disease (RD) is defined as: Any invasive cancer in the breast or axillary lymph nodes in the surgical specimen.
Time Frame: 20 weeks
Population: For ER-negative cancers, the maximum sample size was set to n = 25 and the regimen would be considered of interest if > 20 patients achieve pCR. For ER-positive patients, the maximum sample size for the ER-positive cohort was set to 39 and the regimen would be considered of interest in this subgroup if > 23 patients achieve pCR.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Chemo Plus Pertuzumab,Trastuzumab
Number analyzed (Participants) | 48
proportion of participants
  HR Positive: number analyzed (Participants) | 23
  HR Positive | .26 [.13 to .46]
  HR Negative: number analyzed (Participants) | 25
  HR Negative | .80 [.60 to .91]

2. Secondary Outcome: Cardiac Safety
Description: To assess the safety of the regimen, cardiac safety was measured by rates of clinically symptomatic congestive heart failure, asymptomatic decrease in LVEF >10%, and decrease of LVEF below normal level. This was assessed up to 1 year following surgery.
Time Frame: Up to 1 year post surgery
Population: All patients are assessed in each arm.
Measure: Count of Participants; unit: Participants
Groups:
- Chemo Plus Pertuzumab,Trastuzumab-symptomatic Congestive Heart; Chemo Plus Pertuzumab,Trastuzumab-asympomatic Decrease in LVEF; Chemo Plus Pertuzumab,Trastuzumab-LVEF Below Normal Level: During weeks 1-12, patients will receive pertuzumab, trastuzumab, and paclitaxel at the same time; during weeks 13-24 patients will receive pertuzumab and trastuzumab at the same time with 5-fluorouracil, epirubicin, and cyclophosphamide (FEC).
  Pertuzumab: First dose is 840mg, maintenance dose is 420mg. Pertuzumab will be administered once every 3 weeks for 24 weeks (8 doses total)
  Trastuzumab: For weeks 1-12, first dose is 4 mg/kg, maintenance dose is 2 mg/kg administered every week (12 doses total).
  For weeks 13-24, dose is 6mg/kg administered every 3 weeks (4 doses total).
  Paclitaxel: Administered at 80mg/m2 every week from week 1 to 12 (12 doses total).
  5-fluorouracil: Administered at 500 mg/m2 for every 3 weeks during weeks 13-24 (4 doses total).
  Epirubicin: Administered at 75mg/m2 every 3 weeks during weeks 13-24 (4 doses total).
  Cyclophosphamide: Administered at 500mg/m2 for every 3 weeks during weeks 13-24 (4 doses total).
Arm/Group | Chemo Plus Pertuzumab,Trastuzumab-symptomatic Congestive Heart | Chemo Plus Pertuzumab,Trastuzumab-asympomatic Decrease in LVEF | Chemo Plus Pertuzumab,Trastuzumab-LVEF Below Normal Level
Number analyzed (Participants) | 50 | 50 | 50
Participants | 0 | 14 | 1

3. Secondary Outcome: Count of Patients With Clinical Response
Description: To assess clinical response according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, the number of patients are presented with a clinical response.
Time Frame: Up to 28 weeks
Population: All patients are assessed by HR-positive or HR-negative status.
Measure: Count of Participants; unit: Participants
Groups:
- Chemo Plus Pertuzumab,Trastuzumab HR-positive; Chemo Plus Pertuzumab,Trastuzumab HR-negative: During weeks 1-12, patients will receive pertuzumab, trastuzumab, and paclitaxel at the same time; during weeks 13-24 patients will receive pertuzumab and trastuzumab at the same time with 5-fluorouracil, epirubicin, and cyclophosphamide (FEC).
  Pertuzumab: First dose is 840mg, maintenance dose is 420mg. Pertuzumab will be administered once every 3 weeks for 24 weeks (8 doses total)
  Trastuzumab: For weeks 1-12, first dose is 4 mg/kg, maintenance dose is 2 mg/kg administered every week (12 doses total).
  For weeks 13-24, dose is 6mg/kg administered every 3 weeks (4 doses total).
  Paclitaxel: Administered at 80mg/m2 every week from week 1 to 12 (12 doses total).
  5-fluorouracil: Administered at 500 mg/m2 for every 3 weeks during weeks 13-24 (4 doses total).
  Epirubicin: Administered at 75mg/m2 every 3 weeks during weeks 13-24 (4 doses total).
  Cyclophosphamide: Administered at 500mg/m2 for every 3 weeks during weeks 13-24 (4 doses total).
Arm/Group | Chemo Plus Pertuzumab,Trastuzumab HR-positive | Chemo Plus Pertuzumab,Trastuzumab HR-negative
Number analyzed (Participants) | 23 | 25
Participants | 6 | 20

4. Secondary Outcome: Residual Cancer Burden Score
Description: To assess cancer burben, the Residual Cancer Burden (RCB) score was used. This score has a range of 0 - III, where III (3) is the worst level of burden.
Time Frame: Up to 28 weeks
Population: Total participants that were analyzed for this score (n=43).
Measure: Count of Participants; unit: Participants
Arm/Group | Chemo Plus Pertuzumab,Trastuzumab
Number analyzed (Participants) | 43
Participants
  RCB = 0 | 28
  RCB = I (1) | 5
  RCB = II (2) | 4
  RCB = III (3) | 4

ADVERSE EVENTS:
Time Frame: Up to 28 weeks.
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational medicinal product (IMP) or other protocol-imposed intervention, regardless of attribution.
  This includes the following; AEs not previously observed in the subject that emerge during the protocol, specified AE reporting period. Complications that occur as a result of protocol-mandated interventions (e.g., invasive procedures such as cardiac catheterizations).
Arm/Group | Chemo Plus Pertuzumab,Trastuzumab
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 6/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemo Plus Pertuzumab,Trastuzumab (N=50)
Catheter related infection (Infections and infestations) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (1) — event related to surgery complications
Suicidal ideation (Psychiatric disorders) | 1 (1) — Underlying condition of bi polar disorder
Flu like symptoms (General disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemo Plus Pertuzumab,Trastuzumab (N=50)
Anemia (Blood and lymphatic system disorders) | 36 (65)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Palpitations (Cardiac disorders) | 3 (5)
Blurred vision (Eye disorders) | 5 (5)
Watering eyes (Eye disorders) | 12 (13)
Abdominal pain (Gastrointestinal disorders) | 10 (12)
Constipation (Gastrointestinal disorders) | 14 (15)
Diarrhea (Gastrointestinal disorders) | 45 (110)
Dry mouth (Gastrointestinal disorders) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 7 (8)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 10 (12)
Mucositis oral (Gastrointestinal disorders) | 19 (33)
Nausea (Gastrointestinal disorders) | 41 (67)
Stomach pain (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 13 (18)
Edema limbs (General disorders) | 8 (10)
Fatigue (General disorders) | 43 (59)
Infusion related reaction (General disorders) | 3 (4)
Pain (General disorders) | 27 (49)
Allergic reaction (Immune system disorders) | 4 (5)
Nail infection (Infections and infestations) | 6 (6)
Skin infection (Infections and infestations) | 4 (4)
Upper respiratory infection (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 6 (6)
Alanine aminotransferase increased (Investigations) | 27 (52)
Alkaline phosphatase increased (Investigations) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 16 (20)
Neutrophil count decreased (Investigations) | 13 (21)
Weight loss (Investigations) | 4 (4)
White blood cell decreased (Investigations) | 21 (47)
Anorexia (Metabolism and nutrition disorders) | 5 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (13)
Hypokalemia (Metabolism and nutrition disorders) | 10 (19)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Dizziness (Nervous system disorders) | 10 (12)
Dysgeusia (Nervous system disorders) | 10 (11)
Headache (Nervous system disorders) | 16 (20)
Paresthesia (Nervous system disorders) | 4 (5)
Peripheral motor neuropathy (Nervous system disorders) | 7 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 25 (34)
Anxiety (Psychiatric disorders) | 8 (10)
Insomnia (Psychiatric disorders) | 18 (21)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 4 (6)
Breast pain (Reproductive system and breast disorders) | 5 (6)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 19 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 35 (40)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 38 (50)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8)
Nail discoloration (Skin and subcutaneous tissue disorders) | 18 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 19 (24)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 21 (24)
Scalp pain (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (5)
Flushing (Vascular disorders) | 3 (3)
Hot flashes (Vascular disorders) | 20 (22)
Hypertension (Vascular disorders) | 7 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT01855828/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT01855828/Prot_SAP_001.pdf